CLINICAL TRIAL: NCT03413046
Title: The Effect of Chemotherapy on Regulatory T Cells in Children With Acute Lymphoblastic Leukemia
Brief Title: The Effect of Chemotherapy on Regulatory T Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara Children's Health and Diseases Hematology and Oncology Training and Research Hospital (Other Government)
Collaborators: Turkish Society of Hematology (Other)
Responsible Party: Principal Investigator, Tekin Aksu, Principal Investigator, Ankara Children's Health and Diseases Hematology and Oncology Training and Research Hospital
Other Study IDs: 2017-6
Record Dates: First submitted 2017-12-21; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Pre B ALL; Regulatory T Cell
Keywords: Regulatory T cell; Acute lymphoblastic leukemia; Minimal residual disease
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALL: 30 children with a recent diagnosis of PreB ALL
  Interventions: Diagnostic Test: Peripheral and bone marrow sampling
- Control: 30 healthy children
  Interventions: Diagnostic Test: Peripheral and bone marrow sampling

INTERVENTIONS:
Diagnostic Test: Peripheral and bone marrow sampling — We obtained blood from peripheral and bone marrow sampling. Then we analyze Treg population and Treg related cytokines with flow cytometry and ELISA methods.

SUMMARY:
The investigators aimed to study the effect of chemotherapy on regulatory T cells (Tregs) in children with precursor B (PreB) acute lymphoblastic leukemia (ALL) at 15 and 33 days of malignity directed therapy. The investigators will analyze peripheral and bone marrow blood samples of the participants, obtained at diagnosis, 15 and 33 days of treatment, about Treg / non Treg cells and interleukin (IL)-2, IL-6, IL-10, and transforming growth factor (TGF) beta levels. By this means, investigators will search response to chemotherapy. Also, investigators will analyze correlation between Treg population-Treg related cytokines with demographic, clinical and laboratory findings of the participants with ALL at these certain time points. Additionally, the investigators will compare Treg population and minimal residual disease at 15-33 days of malignity directed therapy. Also investigators will compare these Treg-Treg related cytokines obtained from the participants with ALL and a healthy children control group whom are voluntary donors for bone marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1-18 years
* Recent PreB ALL diagnosis

Exclusion Criteria:

* Children under 1 or over 18 years
* Underlying disease e.g. immune deficiency, germline mutations or diseases
* Tcell ALL or acute myeloid leukemia (AML) patients

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patients diagnosed with PreB ALL in a hematology clinic. Healthy children whom are volunraty bone marrow donors.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in number of regulatory T-cells at 15 and 33th day during chemotherapy | Baseline, 15 and 33th day
  The number of regulatory T-cells is measured in fresh peripheral and bone marrow blood by flow cytometry.

SECONDARY OUTCOMES:
Change from baseline IL-2, IL-6, IL-10, and TGF-beta levels at 15 and 33th day during chemotherapy | Baseline, 15 and 33th day
  IL-2, IL-6, IL-10, and TGF-beta levels are measured in frozen peripheral and bone marrow blood by ELISA.

IPD SHARING:
Plan to Share IPD: Yes